CLINICAL TRIAL: NCT03816371
Title: The Effects of Different Degrees of Head-of-bed Elevation on the Respiratory Pattern and Drainage Following Thyroidectomy: A Randomized Controlled Trial
Brief Title: The Effects of Different Degrees of Head-of-bed Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serpil Yüksel, Assistant Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3029
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Surgery; Thyroid; Nursing Caries
Keywords: thyroidectomy; head-of-bed elevation; supine position; respiratory pattern; amount of drainage; peripheral oxygen saturation
MeSH Terms: conditions — Thyroid Diseases; Deception

STUDY DESIGN:
Intervention Model Description: This study was conducted as a prospective, single-center, parallel, three arm (1:1:1), randomized controlled trial at the Endocrine Surgery Clinic of a university hospital in Turkey.
Who Masked: Participant
Masking Description: Group allocation was concealed using individual sealed opaque envelopes that were numbered in sequential order. As individuals were enrolled in the study, the next envelope in the sequence was extracted and the participant was assigned to the groups accordingly. All the researchers except for the clinical nurse who positioned the patients according to randomization list and patients were blinded from group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- supine 0 degree head-of-bed elevation (Active Comparator): 0 degree head-of-bed elevation was arranged as soon as the patient was admitted to the bed following thyroidectomy.
  Interventions: Other: Head-of-bed elevation
- 30 degree head-of-bed elevation (Experimental): 30 degree head-of-bed elevation was arranged as soon as the patient was admitted to the bed following thyroidectomy.
  Interventions: Other: Head-of-bed elevation
- 45 degree head-of-bed elevation (Experimental): 45 degree head-of-bed elevation was arranged as soon as the patient was admitted to the bed following thyroidectomy.
  Interventions: Other: Head-of-bed elevation

INTERVENTIONS:
Other: Head-of-bed elevation — Respiratory pattern including respiratory rate, peripheral oxygen saturation and dyspnea, and drainage including amount of drainage and hematoma formation of all patients were evaluated at 1st, 2nd, 3rd, and 4th hours after positions.

SUMMARY:
The patient's position is important for ensuring patient comfort and preventing complications after thyroidectomy. This study was carried out to determine the effects of different degrees of head-of-bed elevation on the respiratory pattern and drainage following thyroidectomy and to provide suggestions for evidence-based clinical practice.

DETAILED DESCRIPTION:
Thyroidectomy is a safe surgical procedure commonly used for the treatment of benign or malignant tumors, multinodular goiter and Graves disease. However, because of the rich vascular structure of the thyroid gland, serious complications including hemorrhage, hematoma and hematoma-related dyspnea can develop after thyroidectomy. The American Thyroid Association also suggested to keep the patient in a head-up at 45°-Fowler's position in the post anesthesia care unit following thyroidectomy to prevent hematoma formation on the incision site by facilitating venous return from the head and neck. The mentioned guideline does not offer any recommendations regarding the position that should be given to the patients at surgical clinic after thyroidectomy. Therefore, this study aimed to identify the effects of different degrees of head-of-bed elevation on respiratory pattern including respiratory rate, peripheral oxygen saturation and dyspnea, and drainage including amount of drainage and hematoma formation.

ELIGIBILITY:
Inclusion Criteria: The eligible participants were those

* who were not using anticoagulants,
* whose coagulation tests were normal,
* who had hemovac drains inserted during thyroidectomy,
* who had no contraindication to positioning (e.g., heart failure, chronic obstructive pulmonary disease, dyspnea before surgery and respiratory complications in the post-anesthesia care unit),
* who could tolerate positioning, and who volunteered to participate and signed the informed consent form

Exclusion Criteria:The participants excluded from the study;

* who were using anticoagulants,
* whose coagulation tests were abnormal,
* who had hemovac drains inserted during thyroidectomy,
* hemovac drains removed in the post-anesthesia care unit following thyroidectomy,
* who did not tolerate positioning and who refused to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Respiration rate | Every hour during four hours
  Number of breaths per minute. It is counted for one minute.
Peripheral oxygen saturation | Every hour during four hours
  This oxygen saturation level is used to estimate arterial blood saturation and refers to the amount of oxygenated haemoglobin in the blood. It is measured by an indirect device using non-invasive method.
Amount of drainage | Every hour during four hours
  Drainage is the accumulation of blood in the drain suction bottle. The symptoms including red drainage and drainage more than 150 ml per hour in the suction bottle are defined as bleeding.The drain in the suction bottle is recorded hourly.

SECONDARY OUTCOMES:
Dyspnea | Every hour during four hours
  Shortness of breath (dyspnea) is defined a subjective experience by individuals who complain of unpleasant or uncomfortable respiratory sensations. It is evaluated by patient expression and various instruments.
Hematoma formation | Every hour during four hours
  Hematoma is localized swelling that is filled with blood caused by a break in the wall of a blood vessel. It is evaluated by monitoring warning signs such as progressive neck swelling, hypoxia, tachycardia, dyspnea and stridor.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Yüksel, PhD, Principal Investigator — Necmettin Erbakan University

IPD SHARING:
Plan to Share IPD: No